CLINICAL TRIAL: NCT02501070
Title: Impact of Implantation of PROGALIAM Network (Galician Program of Care in Acute Myocardial Infarction) in Cardiovascular Health in the Northern Area of Galicia.
Brief Title: Impact on Public HEalth of a Network in Acute Myocardial Infarction Care
Acronym: iPHENAMIC
Status: Completed | Type: Observational
Sponsor: Complexo Hospitalario Universitario de A Coruña (Other)
Collaborators: Hospital Universitario Lucus Augusti (Other); Hospital Arquitecto Marcide (Other)
Responsible Party: Principal Investigator, Guillermo Aldama, Interventional Cardiologist, Complexo Hospitalario Universitario de A Coruña
Other Study IDs: D5130C00091
Record Dates: First submitted 2015-07-09; First posted 2015-07-17 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome
Keywords: Percutaneous Coronary Intervention; Angioplasty; Stent; Community Networks
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-PROGALIAM: Patients treated for myocardial infarction before the implementation of the network for acute myocardial infarction care (2001 to 2005).
- PROGALIAM: Patients treated for myocardial infarction after the implementation of the network for acute myocardial infarction care (2005 to 2011).

SUMMARY:
This is a multicenter retrospective observational study with STEMI (ST Elevation Myocardial Infarction) patients who have been treated in the northern Galician Hospitals. The study tries to verify if the implantation of the PROGALIAM (Galician Assistance Program Acute Myocardial Infarction) has supposed a progress in the quality and expectancy of life of AMI patients in the north area of Galicia.

The study will recruit STEMI patients according to the third consensus definition of myocardial infarction type I.

It will include all patients who meet these criteria regardless of other demographic or clinical circumstances. There is not exclusion criteria defined for this population.

DETAILED DESCRIPTION:
* Study Hypothesis This study tries to verify if the implantation of the PROGALIAM has supposed a progress in the quality and expectancy of life of AMI patients in the north area of Galicia.
* Objectives.

The study presents the following objectives:

Primary Objectives:

To compare morbidity rates between pre and post-PROGALIAM periods in major adverse cardiac events. The outcome to study is a composite of death, reinfarction, heart failure and major bleeding at 30 days, one year and long term follow-up.

Secondary Objectives To compare Pre and post PROGALIAM periods regarding;

1. Overall mortality at 30 days, one year and long term follow up. 2. Reinfarction at 30 days, one year and long term follow up. 3. Heart failure incidence at 30 days, one year and long term follow up 4. Hospital major bleeding and at 30 days. 5. Hospital Vascular complications and at 30 days. 6. Heart failure functional Class at 30 days, one year and long term follow up.

* Study Design This is a multicenter retrospective observational study with STEMI patients who have been treated in the northern Galician Hospitals.

  1. Pre-PROGALIAM period: January 2001- May 2005
  2. Post-PROGALIAM period: June 2005- December 2011
* Rational for Sample size Sample size will be constituted by all STEMI cases occurred in both timeframes described above.

According to data obtained in MASCARA register where approximately 38% of ACS patients present ST segment elevation, the estimated sample size would therefore be about 6100 patients.

*Inclusion, Exclusion Criteria and rational The study will recruit STEMI patients according to the third consensus definition of myocardial infarction type I. It was recently published.

It will include all patients who meet these criteria regardless of other demographic or clinical circumstances. There is not exclusion criteria defined for this population.

*Statistical analysis Categorical variables will be presented in percentage, calculated from the whole valid information. The CI will be of 95 %. Quantitative variables will be presented as mean ± standard deviation or median (interquartile range) according to a normal underlying distribution or not. Initially a univariate analysis will be done.

The comparison of quantitative variables means will be done by student´s t-test in case of normality or by nonparametric tests in the opposite case. Categorical variables will be analyzed by the Chi square test. Survival will be analyzed by Kaplan-Meier curves. The comparison between pre and post PROGALIAM curves will be done by a log-rank test. A p <0.05 will be considered statistically significant for two-tailed tests.

Also there are plans to carry out a multivariate analysis. There will be a quantification of the adjusted effect on mortality due to the introduction of PROGALIAM by a Cox Proportional Hazards model. It will be defined the best model to predict this adjusted event by independent variables which can demonstrate an impact on death outcome in the univariate model and by those independent variables in which significant differences are observed between the pre and post PROGALIAM population. The investigators will verify if the implementation of the PROGALIAM is an independent predictor of survival and the impact that generates in the model.

A p <0.05 result will be considered statistically significant in a two-tailed test.

To carry out these analyses it will be necessary to have statistical software like SPSS and/or SAS.

ELIGIBILITY:
Inclusion Criteria:

* All patients suffering STEMI (ST segment Elevation Myocardial Infarction) treated at Northern Galician Network of Acute Myocardial Infarction

Exclusion Criteria:

* No exclusion Criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will gather patients with STEMI (ST segment Elevation Myocardial Infarction) according to the third consensus definition of myocardial infarction treated at Northern Galician Network of Acute Myocardial Infarction.
Sampling Method: Non-Probability Sample
Enrollment: 5937 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Death Pre vs Post PROGALIAM implantation (measured from medical records) | 30 days
  A composite of total death and cardiovascular death
MACE Death Pre vs Post PROGALIAM implantation (Mayor Adverse Cardiovascular Events) (measured from medical records) | 30 days
  A composite of death, reinfarction, heart failure and bleeding
Death Pre vs Post PROGALIAM implantation (measured from medical records) | one year
  A composite of total death and cardiovascular death
MACE Death Pre vs Post PROGALIAM implantation (Mayor Adverse Cardiovascular Events) (measured from medical records) | one year
  A composite of death, reinfarction, heart failure and bleeding

SECONDARY OUTCOMES:
Overall mortality Death Pre vs Post PROGALIAM implantation (measured from medical records) | 30 days, One year
Reinfarction Death Pre vs Post PROGALIAM implantation (measured from medical records) | 30 days, one year
Hospital Mayor bleeding Death Pre vs Post PROGALIAM implantation (measured from medical records) | 30 days
Vascular Complications Death Pre vs Post PROGALIAM implantation (measured from medical records) | 30 days
Heart failure Death Pre vs Post PROGALIAM implantation (measured from medical records) | 30 days, one year

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Aldama, M.D., Study Director — Hospital Universitario de A Coruña; Melisa Santás, M.D., Principal Investigator — Hospital Universitario Lucus Augusti; Manuel Lopez, M.D., Principal Investigator — Hospital Arquitecto Marcide
Locations (1):
- Hospital Universitario de A Coruña, A Coruña, Spain

REFERENCES:
- [Result] Widimsky P, Wijns W, Fajadet J, de Belder M, Knot J, Aaberge L, Andrikopoulos G, Baz JA, Betriu A, Claeys M, Danchin N, Djambazov S, Erne P, Hartikainen J, Huber K, Kala P, Klinceva M, Kristensen SD, Ludman P, Ferre JM, Merkely B, Milicic D, Morais J, Noc M, Opolski G, Ostojic M, Radovanovic D, De Servi S, Stenestrand U, Studencan M, Tubaro M, Vasiljevic Z, Weidinger F, Witkowski A, Zeymer U; European Association for Percutaneous Cardiovascular Interventions. Reperfusion therapy for ST elevation acute myocardial infarction in Europe: description of the current situation in 30 countries. Eur Heart J. 2010 Apr;31(8):943-57. doi: 10.1093/eurheartj/ehp492. Epub 2009 Nov 19. PMID 19933242
- [Result] Widimsky P, Zelizko M, Jansky P, Tousek F, Holm F, Aschermann M; CZECH investigators. The incidence, treatment strategies and outcomes of acute coronary syndromes in the "reperfusion network" of different hospital types in the Czech Republic: results of the Czech evaluation of acute coronary syndromes in hospitalized patients (CZECH) registry. Int J Cardiol. 2007 Jul 10;119(2):212-9. doi: 10.1016/j.ijcard.2007.02.036. Epub 2007 Apr 18. PMID 17442424
- [Result] McManus DD, Gore J, Yarzebski J, Spencer F, Lessard D, Goldberg RJ. Recent trends in the incidence, treatment, and outcomes of patients with STEMI and NSTEMI. Am J Med. 2011 Jan;124(1):40-7. doi: 10.1016/j.amjmed.2010.07.023. PMID 21187184
- [Result] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Result] Mandelzweig L, Battler A, Boyko V, Bueno H, Danchin N, Filippatos G, Gitt A, Hasdai D, Hasin Y, Marrugat J, Van de Werf F, Wallentin L, Behar S; Euro Heart Survey Investigators. The second Euro Heart Survey on acute coronary syndromes: Characteristics, treatment, and outcome of patients with ACS in Europe and the Mediterranean Basin in 2004. Eur Heart J. 2006 Oct;27(19):2285-93. doi: 10.1093/eurheartj/ehl196. Epub 2006 Aug 14. PMID 16908490
- [Result] Jernberg T, Johanson P, Held C, Svennblad B, Lindback J, Wallentin L; SWEDEHEART/RIKS-HIA. Association between adoption of evidence-based treatment and survival for patients with ST-elevation myocardial infarction. JAMA. 2011 Apr 27;305(16):1677-84. doi: 10.1001/jama.2011.522. PMID 21521849
- [Result] Marrugat J, Elosua R, Marti H. [Epidemiology of ischaemic heart disease in Spain: estimation of the number of cases and trends from 1997 to 2005]. Rev Esp Cardiol. 2002 Apr;55(4):337-46. doi: 10.1016/s0300-8932(02)76611-6. Spanish. PMID 11975899
- [Result] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Result] Mamas MA, Ratib K, Routledge H, Fath-Ordoubadi F, Neyses L, Louvard Y, Fraser DG, Nolan J. Influence of access site selection on PCI-related adverse events in patients with STEMI: meta-analysis of randomised controlled trials. Heart. 2012 Feb;98(4):303-11. doi: 10.1136/heartjnl-2011-300558. Epub 2011 Dec 6. PMID 22147900
- [Result] Estevez-Loureiro R, Calvino-Santos R, Vazquez JM, Barge-Caballero E, Salgado-Fernandez J, Pineiro M, Freire-Tellado M, Varela-Portas J, Martinez L, Gomez S, Rodriguez JA, Vazquez N, Castro-Beiras A. Safety and feasibility of returning patients early to their originating centers after transfer for primary percutaneous coronary intervention. Rev Esp Cardiol. 2009 Dec;62(12):1356-64. doi: 10.1016/s1885-5857(09)73529-7. PMID 20038401
- [Result] Barge-Caballero E, Vazquez-Rodriguez JM, Estevez-Loureiro R, Calvino-Santos R, Salgado-Fernandez J, Aldama-Lopez G, Pinon-Esteban P, Flores-Rios X, Campo-Perez R, Rodriguez-Fernandez JA, Lomban-Villanueva JA, Mesias-Prego A, Gutierrez-Cortes JM, Gonzalez-Juanatey C, Portela C, Iglesias-Vazquez A, Varela-Portas Marino J, Vazquez-Gonzalez N, Castro-Beiras A. Primary angioplasty in Northern Galicia: care changes and results following implementation of the PROGALIAM protocol. Rev Esp Cardiol (Engl Ed). 2012 Apr;65(4):341-9. doi: 10.1016/j.recesp.2011.11.003. Epub 2012 Feb 10. PMID 22325936
- [Result] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Result] Ferreira-Gonzalez I, Permanyer-Miralda G, Marrugat J, Heras M, Cunat J, Civeira E, Aros F, Rodriguez JJ, Sanchez PL, Bueno H; MASCARA study research team. MASCARA (Manejo del Sindrome Coronario Agudo. Registro Actualizado) study. General findings. Rev Esp Cardiol. 2008 Aug;61(8):803-16. English, Spanish. PMID 18684363
- [Derived] Aldama G, Lopez M, Santas M, Flores X, Pinon P, Salgado J, Calvino R, Vazquez N, Mesias A, Gonzalez-Juanatey C, Muniz J, Vazquez JM. Impact on mortality after implementation of a network for ST-segment elevation myocardial infarction care. The IPHENAMIC study. Rev Esp Cardiol (Engl Ed). 2020 Aug;73(8):632-642. doi: 10.1016/j.rec.2019.09.031. Epub 2020 Feb 1. English, Spanish. PMID 32014432